### ORI IRB# 00000278

Protocol Version 11/06/2018

Official Title: Talk STEM Familia: A Language Acquisition Smart Speaker-Based App to Improve English Language Acquisition And Family Engagement and Promote Long-Term Educational and Health Outcomes Among First- and Second-Generation Latino Families

Principal Investigators: Jessie Marquez, Patricia Vadasy, Ph.D.

Oregon Research Behavioral Intervention Strategies, Inc. dba Influents Innovations

Award No. R43MD013619 - 01

Final Version Dated: 11/06/2018

### **Informed Consent for Talk STEM Familia Participation**

You and your 4<sup>th</sup>/5<sup>th</sup> grade child are invited to participate in a research study to test Talk STEM Familia, an Alexa skill (app) that helps families support their child's school success. Talk STEM Familia offers lessons and practice in the vocabulary words that support success in STEM (science, technology, engineering, and math).

The Talk STEM Familia study is funded by the National Institute of Minority Health and Health Disparities.

The project is led by Jessie Marquez and Patricia Vadasy, Ph.D. of Influents Innovations in Eugene, OR.

Please read this form and ask any questions you might have before agreeing to participate in this study.

### If You Decide to Participate, You will be Asked to:

- Attend a 1.5 hour group meeting with your child in [month] at a local school or community center.
- Fill out forms with questions on demographics, parenting, and helping your child with school work.
- Provide permission for your child to fill out questionnaires about how he/she feels about school and what kind of help your childwould like at home.
- Receive an Alexa Echo Dot with the Talk STEM skill (app) and learn how to use the app's lessons, games, and activities.
- We will set up an account for you with Amazon so you can use the Alexa Echo Dot. You can keep the Echo Dot after the study is over.
- For the next 6 weeks, receive 3 texts each week reminding you to use Talk STEM with your child for approximately 30 minutes a week, at your convenience.
- At the end of the 6 weeks, attend a 2<sup>nd</sup> group meeting to complete a 2<sup>nd</sup> set of questionnaires. These questionnaires will be similar to the first. In addition we will ask you and your child whether Talk STEM is useful, engaging, and meets family needs.
- At the 2<sup>nd</sup> group meeting, parents will receive \$100. Students, with parent permission, will receive \$25.

# Risks and What Will Be Done to Reduce the Risks

Here are some risks involved for you and your child as participants:

- 1. We will collect some personal information from you and your child. It is possible that someone who is not authorized might see it. We will take these precautions to prevent unauthorized access to the information you give us:
  - a. Any information you or your child give us will be kept strictly confidential. We will keep all information in a locked file. We will remove all names from all the information we get (except this consent form). An ID # will be assigned to the information you give us, and only authorized staff will have access to the locked file that links your name to your ID#.
- 2. Some mass market publications have raised questions concerning the privacy risks associated with smart speaker devices, like the Amazon Echo Dot.
  - a. Amazon appears to take this concern seriously and provides clear visual cues when the device is in a state to capture and send audio to Alexa's back-end infrastructure. Users can also disable the microphone on the device and there are visual cues to indicate that the device is in this state. When an Alexa device is in an active state (microphone enabled), it is listening for the "wake" word (typically, "Alexa") which communicates a user's intent to engage with the device and service. This detection occurs without sending data outside of the device. Audio data is not sent to the cloud until the device detects the wake word to mitigate concerns that

2

Alexa devices are recording indiscriminately. There is no mechanism to remotely trigger recording on Alexa devices independent of local user action.

The Amazon account we set up for you will not have your name on it. We use a number instead.

- 3. You and/or your child might feel uncomfortable if you are unsure about how to answer questions on the questionnaires. We will translate and explain the questions to help you.
- 4. We have a Certificate of Confidentiality, a legal assurance from the federal government that will help us protect your privacy even if the records are subpoenaed. We will not give information to anyone unless you provide a signed release telling us to do so, or unless we have reason to suspect: 1) abuse, neglect, or endangerment of a child or elder; 2) or that anyone is in immediate danger of seriously hurting himself/herself or someone else. In these situations, we may have to make a report to the appropriate authorities.
  - a. If the U. S. Department of Health and Human Services (DHHS) audits our research project, they can have access to information about you. However, they cannot report it to the police or use it for any reason besides the audit.

## **Security**

We collect names, email addresses, mailing addresses, and phone numbers to communicate with you about the study. This information is not stored or associated with the information collected from the surveys. A small amount of email communication is used by the research assistant to schedule and follow up with families.

Communication between the Echo Dot and the Cloud is encrypted. This means that when you speak to the Alexa dot, the speech is coded to make it difficult for someone to access it without permission. After the speech is transmitted to Amazon, the speech remains coded.

Certain unidentifiable data is kept by Amazon to improve the quality of their speech recognition programs. Other data is stored in the password protected account of the user. In this study, the research project staff will manage and own the accounts and will have access to skill usage data within the account. Since the account will be unidentifiable, research staff will not be able to link this data to specific family identifiers. Finally, other data will be stored in the skill's (research project) database. This data will be basic elements such as percentage correct, time spent using the skill, progress, and how often a word was practiced.

#### Benefits to You and Your Child for Participation

You and your child could enjoy learning new vocabulary words and using them to talk about school and home interests. You and your child could enjoy being a part of research that supports the educational and health outcomes of others.

# Your Right to Withdraw from the Study

Your participation is completely voluntary. If you decide not to participate it will not affect school benefits you might otherwise receive. If you decide to participate, you can stop participating any time without penalty.

# **Request for more information**

If you have questions about the research at any time, or if you have a visual or other impairment and require this material in another format, please call: Natasha Compton, Research Assistant (541) 484-2123 x2994 1776 Millrace Dr., Eugene, OR 97403. ORI's TDD number is 800-735-2900

If you have questions about your rights as a research subject, call the Office for the Protection of Human Subjects, Oregon Research Institute, (541) 484-2123. ORI's TDD number is 800-735-2900.

You will be given a copy of this form to keep. Your signature below indicates that you:

| (1) | have read and understand the information provided above, |
|-----|----------------------------------------------------------|
| (2) | agree to participate, |
| (3) | consent to your child's participation, |

(4) may withdraw your consent at any time and stop participating at any time without penalty,

(5) may withdraw your consent for your child's participation at any time without penalty to you or your child (6) have received a copy of this consent form.

| Printed Name (of parent) | Your Child's First Name |
|--------------------------|-------------------------|
| Signature (of parent) | Date |

### CHILD AGREEMENT TO PARTICIPATE

We are asking you to take part in our project to test how well the Talk STEM Family program works for students and families. We will ask you to fill out some questionnaires. We will also ask you and your family to use the Talk STEM Familia app on the Echo Dot for about 30 minutes a week for six weeks. You can decide not to participate at any time.

If you would like to fill out the questionnaires and use the Talk STEM Familia app on the Echo Dot with your family, please sign below.

| AGREE | <b>A</b> ) Y | | |
|-----------------------|--------------|------|---|
| REFUSE | | Date | _ |
| Print Child's Name | | | |
| Oh | | | |
| Witness for Child's A | Assent | | |